CLINICAL TRIAL: NCT02296099
Title: The Impact of Liposomal Bupivacaine Administered Following Placement of a Retropubic Suburethral Sling for Stress Urinary Incontinence: a Randomized Placebo-controlled Trial
Brief Title: Trial Liposomal Bupivacaine Following Retropubic Suburethral Sling for Stress Urinary Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-052
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-02

CONDITIONS: Urinary Incontinence, Stress
Keywords: retropubic suburethral sling; stress urinary incontinence; liposomal bupivacaine
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): The placement of the retropublic sling will be placed in routine fashion under general anesthesia. If randomized to liposomal bupivacaine, the standard 20 milliliter (ml) vial (266mg dose) will be diluted with 10ml of preservative-free, sterile normal saline (0.9%) for injection to a reconstituted volume of 30ml. At the completion of the procedure, and at least 20 minutes after the injection of 30ml lidocaine with epinephrine (routine for the surgical procedure), those subjects in the liposomal bupivacaine arm will have the 30ml dilutional volume injected. 10ml will be injected into the vaginal epithelium in the mid-urethral area and 10ml will be injected into each of the trocar paths through the suprapubic incisions bilaterally. An aspiration and moving needle technique will be employed.
  Interventions: Drug: liposomal bupivacaine
- Saline Placebo (Placebo Comparator): The placement of the retropublic sling will be placed in routine fashion under general anesthesia. At the completion of the procedure, and at least 20 minutes after the injection of 30ml lidocaine with epinephrine (routine for the surgical procedure), those subjects in the saline placebo arm will receive 30ml normal saline injected. 10ml will be injected into the vaginal epithelium in the mid-urethral area and 10ml will be injected into each of the trocar paths through the suprapubic incisions bilaterally. An aspiration and moving needle technique will be employed.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: liposomal bupivacaine — Liposomal bupivacaine 20 mL diluted with 10 mL normal saline. Ten mL of solution to be injected into the vaginal epithelium in the mid-urethral area and 10 mL injected into each of the trocar paths through the suprapubic incisions bilaterally.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Placebo — Normal saline 30 mL total injected. Ten mL injected into the vaginal epithelium in the mid-urethral area and 10 mL will be injected into each of the trocar paths through the suprapubic incisions bilaterally.
  Other Names: Normal Saline
  Arms: Saline Placebo

SUMMARY:
The purpose of the study is to determine if the administration of liposomal bupivacaine at the completion of a suburethral sling procedure will result in decreased postoperative pain compared to no injection.

DETAILED DESCRIPTION:
The purpose of the study is to determine if the administration of liposomal bupivacaine at the completion of a suburethral sling procedure will result in decreased postoperative pain compared to no injection. The hypothesis is that administration of liposomal bupivacaine at the completion of retropubic suburethral sling procedure will result in decreased postoperative pain compared to no injection. Although multiple routes for sling placement exist, no difference in pain has been found when comparing obturator verses retropubic suburethral sling. Previous trials have investigated varying formulations of injections along the sling pathway in order to reduce complications such as pain and voiding dysfunction. Local anesthesia along the trocar pathway has shown some improvements in pain. Other techniques, however, have varying results. In 2011, the FDA approved liposomal bupivacaine as a single dose wound infiltration for treatment of postoperative pain following hemorrhoidectomy and bunionectomy. Initial studies demonstrated decreased pain compared to placebo, prolonged release in a bimodal distribution, and greater sensory than motor blockade. Additionally, postoperative benefits such as decreased overall pain, decreased opioid use, and increased time to opioid need were observed. Liposomal bupivacaine may also have the advantage of reducing hospital stays and decreasing overall hospital costs. The side effect profile has similar or improved rates of adverse events compared to traditional bupivacaine, a favorable cardiac profile, and no increased risk of poor wound healing. With such promise, we aim to evaluate the use of liposomal bupivacaine to reduce postoperative pain for the placement of slings to treat stress urinary incontinence. The study will be a blinded randomized controlled trial. Patients randomized to receive liposomal bupivicaine, the standard 20ml vial will be diluted with 1 Oml of saline to a reconstituted volume of 30 ml. Those in the control group will receive 30ml of normal saline injected in the same fashion as the study arm.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than 18 years of age
* Planning for outpatient surgical treatment of stress urinary incontinence with placement of a retropubic suburethral sling under general anesthesia

Exclusion Criteria:

* Pregnant or nursing
* Allergy to bupivacaine
* History of drug/alcohol abuse
* Severe cardiovascular, hepatic, renal disease, or neurological impairment
* Long-acting opioid within 3 days or any opioid use within 24 hours before surgery
* Contraindication to: acetaminophen, oxycodone, and/or non-steroidal anti-inflammatory drugs (NSAID)
* Administration of an investigational drug within 30 days before study
* Chronic pain syndromes
* Daily NSAID/opioid use
* Patients having concomitant procedures or not undergoing general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, MSc, Principal Investigator — TriHealth Inc.
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Placebo: Normal saline 30 mL total injected. Ten mL injected into the vaginal epithelium in the mid-urethral area and 10 mL will be injected into each of the trocar paths through the suprapubic incisions bilaterally.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Started | 57 | 57
Completed | 54 | 55
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Saline Placebo | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11) | 53 (10) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 55 | 109
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 50 | 53 | 103
  Race: African American | 2 | 2 | 4
  Race: Asian | 1 | 0 | 1
  Race: Latina | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Pain in the Morning
Description: A visual analog scale (VAS) will be used to have the patient rate her pain in the morning of postoperative day one. The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
scores on a scale | 9.5 [2 to 33.25] | 27.0 [8 to 48]
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Saline Placebo; The null hypothesis is that there is no difference in the pain scores between the two groups; Test type: Equivalence — The Mann-Whitney U test was utilized; p = 0.014, Wilcoxon (Mann-Whitney) — The p-value was not adjusted for multiple comparisons; There were no adjustments

2. Secondary Outcome: Pain Upon Discharge From Post-anesthesia Care Unit (PACU)
Description: A visual analog scale (VAS) will be used to have the patient rate her pain upon discharge from the PACU. The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
score on a scale | 1.0 [0.0 to 9.0] | 1.0 [0.0 to 10.0]

3. Secondary Outcome: Pain Upon Discharge From Same Day Surgery
Description: A visual analog scale (VAS) will be used to have the patient rate her pain upon discharge from same day surgery. The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
score on a scale | 2.0 [0.0 to 11.25] | 4.0 [0.0 to 22.0]

4. Secondary Outcome: Pain at Four Hours After Discharge Home
Description: A visual analog scale (VAS) will be used to have the patient rate her pain four hours after being discharged home. The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: 1 day, 4 hours after discharge from Same Day Surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
score on a scale | 3.5 [1.0 to 23.25] | 13.0 [3.0 to 42.0]

5. Secondary Outcome: Total Narcotic Consumption
Description: Cumulative consumption postoperative days 1 - 3
Time Frame: Day 1 - 3
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
morphine equivalents | 11.50 (12.92) | 13.39 (8.24)

6. Secondary Outcome: Number of Participants Reporting 'Very Satisfied' at the 1 Week Postoperative Visit
Description: A likert type scale will be used to have the patient rate their satisfaction with pain control at their one week postoperative visit. Count information for those who were very satisfied were provided.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
Participants | 39 | 45

7. Other Pre Specified Outcome: Number of Participants Reporting 'Very Satisfied' at the 2 Week Postoperative Visit
Description: A likert type scale will be used to have the patient rate their satisfaction with pain control at their two week postoperative visit. Count information for those who were very satisfied were provided.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
Participants | 47 | 49

8. Other Pre Specified Outcome: Pain at Bedtime (Current Level of Pain)
Description: Before going to bed each night the patient will record their pain level at that moment using a visual analog scale (VAS). The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
score on a scale | 18.5 [5.0 to 43.25] | 24.0 [9.0 to 46.0]

9. Other Pre Specified Outcome: Pain at Bedtime (Most Intense Pain)
Description: Before going to bed each night the patient will record the most intense pain using a visual analog scale (VAS). The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
score on a scale | 34.5 [7.75 to 64.0] | 34.5 [20.0 to 55.0]

10. Other Pre Specified Outcome: Pain at Bedtime (Average Pain)
Description: Before going to bed each night the patient will record the average level of pain using a visual analog scale (VAS). The VAS scale ranges from 0 to 100 mm. The higher the VAS score the greater the level of pain reported.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Number analyzed (Participants) | 54 | 55
score on a scale | 21.5 [7.0 to 39.5] | 21.5 [12.0 to 40.0]

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 0/57 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes